CLINICAL TRIAL: NCT04371575
Title: Symptomatic Trigeminal Neuralgia Attributed to Multiple Sclerosis - Clinical Characteristics, Neuroanatomical Abnormalities and Treatment Efficacy
Brief Title: Symptomatic Trigeminal Neuralgia Attributed to Multiple Sclerosis - a Prospective Study in 60 Patients
Status: Completed | Type: Observational
Sponsor: Stine Maarbjerg, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Stine Maarbjerg, MD PhD, Post doc, Danish Headache Center
Organization: Danish Headache Center (Other)
Other Study IDs: 010919
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Trigeminal Neuralgia; Multiple Sclerosis; Pain, Neuropathic
MeSH Terms: conditions — Trigeminal Neuralgia; Multiple Sclerosis; Neuralgia | interventions — Carbamazepine; Oxcarbazepine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Carbamazepine — There is no actual intervention as the study is observational. First choice tratment is Carbamzepine and Oxcarbazepine. In medically refractory patients, first choice surgery is microvascular decompression
  Other Names: Oxcarbazepine

SUMMARY:
Clinical characteristics, neuroanatomical findings and efficacy of medical and surgical treatment of symptomatic trigeminal neuralgia - a systematic prospective study of 60 consecutive patients

DETAILED DESCRIPTION:
Background Among patients with TN, approximately 15% has secondary TN caused by another underlying condition such as multiple sclerosis or a tumor. Studies of classical TN patients have shown a strong association between a severe NVC of the trigeminal nerve and the painful side. This association has been less investigated in STN.

There are no previous systemic and prospective studies of the underlying causes, characteristics and treatment response of patients with STN. Most existing studies on STN have various methodological drawbacks as inclusion was not prospective, diagnosis was not consistent with international guidelines, imaging techniques were not adequately advanced at the time of publication and evaluation of treatment efficacy was not performed by evaluators independent of the neurosurgeon.

Aims

1) To describe the clinical characteristics, the neuroanatomical findings using 3.0 Tesla MRI, and the efficacy of medical and surgical treatment in STN

Hypotheses

1. In STN, there is a correlation between demylinating brainstem plaques and presence and degree of neurovascular contact of the trigeminal nerve ipsilateral to the painful side
2. The efficacy of medical and surgical treatment of STN is comparable to the efficacy in patients with classical trigeminal neuralgia

Power calculations Sample size depends on the number of patients in the inclusion period. The estimated number of included patients is at least 60 patients.

Methods Data have been collected prospectively since 2012 based on semi-structured interview forms completed at out-patient visits at the Danish Headache Center. The efficacy of medical and surgical treatment was also documented prospectively by structured interviews. Efficacy of surgical treatment was evaluated by independent assessors.

All patients had a 3.0 Tesla MRI with a special protocol adapted for the trigeminal nerve and the brainstem.

Ethical considerations The treatment of patients with STN will not differ from the usual treatment and decision-taking.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of secondary trigeminal neuralgia attributed to multiple sclerosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical cohort of patients diagnosed with secondary trigeminal neuralgia attributed to multiple sclerosis at the Danish Headache Center
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Demyelinating brainstem plaques and neurovascular contact | 2012-2019
  In STN, there is a correlation between demyelinating brainstem plaques and presence and degree of neurovascular contact of the trigeminal nerve ipsilateral to the painful side

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bendtsen, Dr Med Sci, Principal Investigator — Danish Headache Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noory N, Smilkov EA, Frederiksen JL, Heinskou TB, Andersen ASS, Bendtsen L, Maarbjerg S. Neurovascular contact plays no role in trigeminal neuralgia secondary to multiple sclerosis. Cephalalgia. 2021 Apr;41(5):593-603. doi: 10.1177/0333102420974356. Epub 2020 Nov 28. PMID 33249870